CLINICAL TRIAL: NCT06058390
Title: A Phase 1, Randomized, Open-Label, Parallel Group Study to Evaluate the Relative Bioavailability of Subcutaneous Bepirovirsen When Delivered From a Vial or Prefilled Syringe Fitted With a Safety Syringe Device in Healthy Adult Participants
Brief Title: A Study to Evaluate the Relative Bioavailability of Subcutaneous Bepirovirsen When Delivered From a Vial or Prefilled Syringe Fitted With a Safety Syringe Device in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 219239
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Hepatitis; Viral; Human; Virus Diseases; Bepirovirsen; GSK3228836; 219239; Liver Diseases
MeSH Terms: conditions — Hepatitis B; Hepatitis; Virus Diseases; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bepirovirsen Vial by HCP (Experimental): Participants will receive Bepirovirsen vial administered by Healthcare Professionals (HCP).
  Interventions: Drug: Bepirovirsen
- Bepirovirsen PFS SSD by HCP (Experimental): Participants will receive Bepirovirsen PFS SSD administered by HCP.
  Interventions: Drug: Bepirovirsen
- Bepirovirsen PFS SSD self-administered post-training (Experimental): Participants will receive Bepirovirsen PFS SSD self- administered with training by HCP.
  Interventions: Drug: Bepirovirsen
- Bepirovirsen PFS SSD self-administered without training (Experimental): Participants will receive Bepirovirsen PFS SSD self- administered with no training by HCP.
  Interventions: Drug: Bepirovirsen

INTERVENTIONS:
Drug: Bepirovirsen — Bepirovirsen will be administered.

SUMMARY:
This is an open-label, randomized study to investigate subcutaneous (SC) bepirovirsen when delivered via SC injection from vial or Prefilled syringe fitted with a Safety syringe device (PFS SSD) in healthy adult participants. The aim of this study is to provide relative bioavailability data to support the transition from the vial presentation of bepirovirsen, to a ready-to-use liquid in a PFS SSD when both are given by a health care professional. The study will also assess self-administration using the PFS SDD, and the safety and tolerability of bepirovirsen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by medical evaluation including medical history, physical examination, laboratory tests, electrocardiogram (ECGs) and vital signs.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and protocol.

Exclusion Criteria:

* Past or current medical conditions which, in the judgement of the investigator and Medical Monitor, could jeopardize the integrity of the data derived from that participant or the safety of the participant.
* Abnormal blood pressure as determined by the investigator.
* Positive Hepatitis B virus (HBV), Hepatitis C virus (HCV) or human immunodeficiency virus (HIV) test results.
* Participants with signs or symptoms suggestive of Coronavirus disease 2019 (COVID-19) within 14 days of inpatient admission, or with a positive test for active COVID-19 infection before study start.
* Past, current or intended use of over the counter or prescription medication [including herbal medications]
* Current or prior use of creatine-containing supplements and intended use up to 50 days post-dosing.

Prior use of immunosuppressive drugs within 3 months before dosing or interferon within 12 months before dosing.

* Prior treatment with any oligonucleotide or small interfering ribonucleoside (RNA) siRNA within 12 months before dosing.
* Loss of blood or blood products in excess of 500 millilitre (mL) within any 3-month period during the study.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation in another investigational study in which an investigational intervention (e.g., drug, vaccine, invasive device) was administered within 5-half-lives (if known) or twice the duration of biological effect (if known), whichever is longer, or within the last 90 days (if half-life and duration of biological effect are unknown), before the first dosing day in the current study.
* Current enrolment or past participation in this clinical study.
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Regular alcohol consumption of alcohol within 6 months prior to the study.
* Regular use of known drugs of abuse, including Tetrahydrocannabinol (THC).
* History of sensitivity to bepirovirsen or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor contraindicates their participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Derived] Youssef AS, Shah P, Hu M, Plein H, Roy A, Sharma R, Mole S, Blazejczyk M, Cross W, Spears B, Pak S, Kaur R, Elston R, Theodore D, Hezareh M, Nader A. A Phase 1, Randomized, Open-Label, Parallel Group Study to Evaluate the Relative Bioavailability and Safety of Subcutaneous Bepirovirsen when Delivered from a Vial or Prefilled Syringe Fitted with a Safety Syringe Device in Healthy Adult Participants. Clin Pharmacol Drug Dev. 2025 Oct 14. doi: 10.1002/cpdd.1615. Online ahead of print. PMID 41085094

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 160 participants were enrolled in the study which were randomized in 4 groups. (Enrolled Population: All participants who entered the study [who were randomized or received study intervention or underwent a post-screening procedure]).
Groups:
- Bepirovirsen 300 mg Vial by HCP: Participants received a single dose of Bepirovirsen (GSK3228836) 300 milligrams (mg) (2*150 mg) subcutaneous (SC) injection packaged in a vial, administered by Healthcare Professionals (HCP).
- Bepirovirsen 300 mg PFS SSD by HCP: Participants received a single dose of Bepirovirsen 300 mg (2*150 mg) SC injection packaged in a prefilled syringe (PFS) fitted with a safety syringe device (SSD), administered by HCP.
- Bepirovirsen 300 mg PFS SSD Self-administered Post-training: Participants received a single dose of Bepirovirsen 300 mg (2*150 mg) SC injection packaged in a PFS fitted with a SSD, self-administered with training from HCP. Participants were monitored by HCP during self-administration.
- Bepirovirsen 300 mg PFS SSD Self-administered Without Training: Participants received a single dose of Bepirovirsen 300 mg (2*150 mg) SC injection packaged in a PFS fitted with a SSD, self-administered with no training from HCP. Participants were monitored by HCP during self-administration.
Period: Overall Study
Arm/Group | Bepirovirsen 300 mg Vial by HCP | Bepirovirsen 300 mg PFS SSD by HCP | Bepirovirsen 300 mg PFS SSD Self-administered Post-training | Bepirovirsen 300 mg PFS SSD Self-administered Without Training
Started (Enrolled Population) | 46 | 49 | 32 | 33
Safety Population | 46 | 49 | 32 | 32
Completed | 46 | 49 | 30 | 30
Not Completed | 0 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Participants did not receive any study intervention | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for the Safety Population which included participants who received study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bepirovirsen 300 mg Vial by HCP | Bepirovirsen 300 mg PFS SSD by HCP | Bepirovirsen 300 mg PFS SSD Self-administered Post-training | Bepirovirsen 300 mg PFS SSD Self-administered Without Training | Total
Number analyzed (Participants) | 46 | 49 | 32 | 32 | 159
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 35.7 (9.09) | 36.5 (9.57) | 36.6 (9.35) | 37.5 (9.74) | 36.5 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 15 | 16 | 82
  Male | 20 | 24 | 17 | 16 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The "All Other Races" category (AMERICAN INDIAN OR ALASKA NATIVE, ASIAN, BLACK OR AFRICAN AMERICAN, MIXED RACE, NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER and where 0<n<11) are combined into one category to maintain participant confidentiality and privacy.
  Participants
    WHITE | 25 | 20 | 13 | 18 | 76
    All Other Races | 21 | 29 | 19 | 14 | 83

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Administration of Bepirovirsen Using Vial and PFS by HCP
Description: Blood samples were collected at indicated timepoints for pharmacokinetic analysis of Bepirovirsen. Cmax calculation for this outcome measure is based on changes in model specifications and inclusion of different arms for respective outcome measures. Model includes Randomized Groups (Groups compared), injection site (arm, thigh and abdomen) as categorical covariates and log transformed Baseline weight as continuous covariate. The treatment is a factor in the model and position of a treatment as either test or reference would affect the Cmax values for a particular outcome measure due to differences in how the model accounts for variability and compares group for mean calculation. Pharmacokinetic (PK) Parameter Population included all participants in the PK concentration Population for whom valid and evaluable plasma PK parameters were derived.
Time Frame: Pre-dose (Day 1) and Post-dose (1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, 168 hours, 336 hours, 672 hours, 1008 hours and 1512 hours)
Population: PK parameter population was the analysis set used. Test group in this outcome measure is Bepirovirsen 300 mg PFS SSD by HCP and reference group is Bepirovirsen 300 mg Vial by HCP for this outcome measure. Based on the test and reference, data was analyzed and Cmax values were modelled as described in measure description which vary across different outcome measures.
Measure: Geometric Mean (Standard Error); unit: Nanograms per milliliters (ng/mL)
Arm/Group | Bepirovirsen 300 mg Vial by HCP | Bepirovirsen 300 mg PFS SSD by HCP
Number analyzed (Participants) | 46 | 49
Nanograms per milliliters (ng/mL) | 9954.89 (0.049) | 10163.74 (0.048)
Statistical Analysis 1: Comparison: Bepirovirsen 300 mg Vial by HCP vs Bepirovirsen 300 mg PFS SSD by HCP; Analysis was performed on the natural logarithms using a fixed-effects model; Test type: Other; Geometric mean ratio = 1.02, 90% CI 2-sided [0.91 to 1.14] — Geometric mean is adjusted for covariates: randomized groups (Arms 1 and 2 of this endpoint), injection site (arm, thigh and abdomen) as categorical covariates and log transformed Baseline weight as continuous covariate

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC [0-Inf]) Following Administration of Bepirovirsen Using Vial and PFS by HCP
Description: Blood samples were collected at indicated timepoints for pharmacokinetic analysis of Bepirovirsen. Blood samples were collected at indicated timepoints for PK analysis of Bepirovirsen. AUC(0-inf) calculation for this outcome measure is based on changes in model specifications and inclusion of different arms for respective outcome measures. Model includes Randomized Groups (Groups compared), injection site (arm, thigh and abdomen) as categorical covariates and log transformed Baseline weight as continuous covariate. The treatment is a factor in the model and position of a treatment as either test or reference would affect the AUC(0-inf) values for a particular outcome measure due to differences in how the model accounts for variability and compares group for mean calculation.
Time Frame: as for outcome 1
Population: PK parameter population was the analysis set used. Test group in this outcome measure is Bepirovirsen 300 mg PFS SSD by HCP and reference group is Bepirovirsen 300 mg Vial by HCP for this outcome measure. Based on the test and reference, data was analyzed and AUC(0-inf) values were modelled as described in measure description which vary across different outcome measures.
Measure: Geometric Mean (Standard Error); unit: Hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Bepirovirsen 300 mg Vial by HCP | Bepirovirsen 300 mg PFS SSD by HCP
Number analyzed (Participants) | 46 | 49
Hours*nanogram per milliliter (h*ng/mL) | 112495.66 (0.039) | 118622.59 (0.038)
Statistical Analysis 1: Comparison: Bepirovirsen 300 mg Vial by HCP vs Bepirovirsen 300 mg PFS SSD by HCP; Analysis was performed on the natural logarithms using a fixed-effects model; Test type: Other; Geometric mean ratio = 1.05, 90% CI 2-sided [0.96 to 1.15] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Administration of Bepirovirsen Using PFS SSD by HCP and PFS SSD Self-administered Post-training
Description: Blood samples were collected at indicated timepoints for pharmacokinetic analysis of Bepirovirsen. Cmax calculation for this outcome measure is based on changes in model specifications and inclusion of different arms for respective outcome measures. Model includes Randomized Groups (Groups compared), injection site (arm, thigh and abdomen) as categorical covariates and log transformed Baseline weight as continuous covariate. The treatment is a factor in the model and position of a treatment as either test or reference would affect the Cmax values for a particular outcome measure due to differences in how the model accounts for variability and compares group for mean calculation.
Time Frame: as for outcome 1
Population: PK parameter population was the analysis set used. Test group in this outcome measure is Bepirovirsen 300 mg PFS SSD self-administered post-training and reference group is Bepirovirsen 300 mg PFS SSD by HCP for this outcome measure. Based on the test and reference, data was analyzed and Cmax values were modelled as described in measure description which vary across different outcome measures.
Measure: Geometric Mean (Standard Error); unit: Nanograms per milliliters
Arm/Group | Bepirovirsen 300 mg PFS SSD by HCP | Bepirovirsen 300 mg PFS SSD Self-administered Post-training
Number analyzed (Participants) | 49 | 29
Nanograms per milliliters | 10225.39 (0.050) | 10421.21 (0.067)
Statistical Analysis 1: Comparison: Bepirovirsen 300 mg PFS SSD by HCP vs Bepirovirsen 300 mg PFS SSD Self-administered Post-training; Analysis was performed on the natural logarithms using a fixed-effects model; Test type: Other; Geometric mean ratio = 1.02, 90% CI 2-sided [0.88 to 1.18] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: AUC(0-inf) Following Administration of Bepirovirsen Using PFS SSD by HCP and PFS SSD Self-administered Post-training
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK parameter population was the analysis set used. Test group in this outcome measure is Bepirovirsen 300 mg PFS SSD self-administered post-training and reference group is Bepirovirsen 300 mg PFS SSD by HCP for this outcome measure. Based on the test and reference, data was analyzed and AUC(0-inf) values were modelled as described in measure description which vary across different outcome measures.
Measure: Geometric Mean (Standard Error); unit: Hours*nanograms per milliliters
Arm/Group | Bepirovirsen 300 mg PFS SSD by HCP | Bepirovirsen 300 mg PFS SSD Self-administered Post-training
Number analyzed (Participants) | 49 | 29
Hours*nanograms per milliliters | 120034.02 (0.038) | 117805.29 (0.050)
Statistical Analysis 1: Comparison: Bepirovirsen 300 mg PFS SSD by HCP vs Bepirovirsen 300 mg PFS SSD Self-administered Post-training; Analysis was performed on the natural logarithms using a fixed-effects model; Test type: Other; Geometric mean ratio = 0.98, 90% CI 2-sided [0.88 to 1.09] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Administration of Bepirovirsen Using PFS SSD by HCP and PFS SSD Self-administered Without Training
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK parameter population was the analysis set used. Test group in this outcome measure is Bepirovirsen 300 mg PFS SSD self-administered without training and reference group is Bepirovirsen 300 mg PFS SSD by HCP for this outcome measure. Based on the test and reference, data was analyzed and Cmax values were modelled as described in measure description which vary across different outcome measures.
Measure: Geometric Mean (Standard Error); unit: Nanograms per milliliters
Arm/Group | Bepirovirsen 300 mg PFS SSD by HCP | Bepirovirsen 300 mg PFS SSD Self-administered Without Training
Number analyzed (Participants) | 49 | 29
Nanograms per milliliters | 10007.69 (0.046) | 9896.63 (0.061)
Statistical Analysis 1: Comparison: Bepirovirsen 300 mg PFS SSD by HCP vs Bepirovirsen 300 mg PFS SSD Self-administered Without Training; Analysis was performed on the natural logarithms using a fixed-effects model; Test type: Other; Geometric mean ratio = 0.99, 90% CI 2-sided [0.87 to 1.13] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: AUC(0-Inf) Following Administration of Bepirovirsen Using PFS SSD by HCP and PFS SSD Self-administered Without Training
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK parameter population was the analysis set used. Test group in this outcome measure is Bepirovirsen 300 mg PFS SSD self-administered without training and reference group is Bepirovirsen 300 mg PFS SSD by HCP for this outcome measure. Based on the test and reference, data was analyzed and AUC(0-inf) values were modelled as described in measure description which vary across different outcome measures.
Measure: Geometric Mean (Standard Error); unit: Hours*nanograms per milliliters
Arm/Group | Bepirovirsen 300 mg PFS SSD by HCP | Bepirovirsen 300 mg PFS SSD Self-administered Without Training
Number analyzed (Participants) | 49 | 29
Hours*nanograms per milliliters | 117938.68 (0.037) | 114492.19 (0.049)
Statistical Analysis 1: Comparison: Bepirovirsen 300 mg PFS SSD by HCP vs Bepirovirsen 300 mg PFS SSD Self-administered Without Training; Analysis was performed on the natural logarithms using a fixed-effects model; Test type: Other; Geometric mean ratio = 0.97, 90% CI 2-sided [0.87 to 1.08] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected up to Day 64
Description: All-cause mortality, SAEs and non-SAEs were reported for Safety Population which included participants who received study intervention. One participant from Enrolled Population (N=160) did not receive study intervention, hence was not included in Safety Population (N=159).
Arm/Group | Bepirovirsen 300 mg Vial by HCP | Bepirovirsen 300 mg PFS SSD by HCP | Bepirovirsen 300 mg PFS SSD Self-administered Post-training | Bepirovirsen 300 mg PFS SSD Self-administered Without Training
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/49 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/49 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 45/46 | 43/49 | 32/32 | 30/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bepirovirsen 300 mg Vial by HCP (N=46) | Bepirovirsen 300 mg PFS SSD by HCP (N=49) | Bepirovirsen 300 mg PFS SSD Self-administered Post-training (N=32) | Bepirovirsen 300 mg PFS SSD Self-administered Without Training (N=32)
Injection site erythema (General disorders) | 35 | 37 | 30 | 30
Injection site swelling (General disorders) | 21 | 24 | 14 | 19
Injection site pain (General disorders) | 23 | 22 | 10 | 12
Injection site pruritus (General disorders) | 8 | 11 | 9 | 13
Injection site discolouration (General disorders) | 7 | 5 | 6 | 5
Injection site pallor (General disorders) | 6 | 3 | 5 | 3
Injection site haemorrhage (General disorders) | 5 | 2 | 3 | 1
Injection site bruising (General disorders) | 2 | 3 | 4 | 1
Injection site warmth (General disorders) | 3 | 2 | 2 | 0
Pyrexia (General disorders) | 3 | 2 | 1 | 1
Chills (General disorders) | 2 | 0 | 1 | 2
Injection site inflammation (General disorders) | 1 | 0 | 2 | 0
Injection site nodule (General disorders) | 2 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0
Medical device site dermatitis (General disorders) | 1 | 0 | 1 | 0
Feeling of body temperature change (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Injection site dermatitis (General disorders) | 0 | 0 | 0 | 1
Injection site discomfort (General disorders) | 0 | 1 | 0 | 0
Injection site exfoliation (General disorders) | 0 | 0 | 0 | 1
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 1
Injection site scab (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Vessel puncture site reaction (General disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 12 | 5 | 5 | 7
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1
Presyncope (Nervous system disorders) | 2 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 2 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil percentage increased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract discomfort (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT06058390/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT06058390/SAP_001.pdf